CLINICAL TRIAL: NCT00971425
Title: Immunogenicity and Safety of GSK Biologicals' Pandemic Influenza Candidate Vaccine GSK2340272A
Brief Title: Evaluation of the Immune Response and the Safety of a Pandemic Influenza Candidate Vaccine (H1N1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 113572
Record Dates: First submitted 2009-08-27; First posted 2009-09-03 (Estimated); Results first posted 2011-03-04 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2017-01

CONDITIONS: Influenza
Keywords: influenza infection; GSK Bio's influenza vaccine GSK2340272A
MeSH Terms: conditions — Influenza, Human | interventions — pandemrix; fluarix

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Placebo-Pandemrix-Fluarix Group (Experimental): Subjects received one dose of placebo intramuscularly in the deltoid region of the dominant arm at Day -21, 2 doses of Pandemrix (GSK2340272A) intramuscularly in the deltoid region of the non-dominant arm at Day 0 and Day 21, and 1 dose of Fluarix intramuscularly in the deltoid region of the dominant arm at Day 42.
  Interventions: Biological: Pandemrix (GSK investigational influenza GSK2340272A vaccine); Biological: Fluarix™; Biological: Placebo
- Fluarix-Pandemrix-Placebo Group (Experimental): Subjects received 1 dose of Fluarix intramuscularly in the deltoid region of the dominant arm at Day -21, 2 doses of Pandemrix (GSK2340272A) intramuscularly in the deltoid of the non-dominant arm at Day 0 and 21, and 1 dose of placebo intramuscularly in the deltoid of the non-dominant arm at Day 42.
  Interventions: Biological: Pandemrix (GSK investigational influenza GSK2340272A vaccine); Biological: Fluarix™; Biological: Placebo

INTERVENTIONS:
Biological: Pandemrix (GSK investigational influenza GSK2340272A vaccine) — 2 doses intramuscular injections
Biological: Fluarix™ — 1 dose intramuscular injection
Biological: Placebo — 1 dose intramuscular injection

SUMMARY:
The objective of the study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK2340272A.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 61 years of age or older at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Satisfactory baseline medical assessment by history and physical examination (stable health status with no exclusionary medical or psychiatric conditions). Stable health status is defined as the absence of health event satisfying the definition of a serious adverse event, or a change in an ongoing drug therapy due to therapeutic failure or symptoms of drug toxicity, within one month prior to enrolment.

Exclusion Criteria:

* Previous administration of the 2009 Southern Hemisphere or 2009-2010 Northern Hemisphere influenza vaccine.
* Previous administration of a pandemic influenza vaccine.
* Administration of any vaccine within 30 days before first vaccination.
* Planned administration of a vaccine not foreseen by the study protocol one month (minimum 30 days) after the second vaccination with the GSK2340272A candidate vaccine.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of the study vaccines or planned use during the study period. Potential subjects in the follow-up phase of a prior investigational study may be enrolled if the investigator's judgment is that it will have no effect on safety, reactogenicity, or immunogenicity endpoints in this study, and that it does not violate the protocol requirements of the prior trial.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of an axillary temperature >= 37.5°C, or acute symptoms greater than "mild" severity on the scheduled date of first vaccination. NOTE: The subject may be vaccinated at a later date, provided symptoms have resolved, vaccination occurs within the window specified by the protocol, and all other eligibility criteria continue to be satisfied.
* Diagnosed with cancer, or treatment for cancer, within 3 years.

  * Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
  * Persons with a history of histological-confirmed basal cell carcinoma of the skin successfully treated with local excisions only are eligible and may be enrolled within 3 years of diagnosis, but other histological types of skin cancer require a 3-year untreated and disease-free window as above.
  * Women who are disease free for 3 years or more after the treatment of breast cancer and receiving long-term prophylactic tamoxifen are eligible and may be enrolled.
* Any confirmed or suspected immunosuppressive or immunodeficient condition including history of human immunodeficiency virus (HIV) infection.
* Chronic administration of immunosuppressants or other immune modifying drugs within six months prior to the first vaccination and during the entire study period.
* Receipt of any immunoglobulins and/or any blood products within 3 months preceding the first vaccination or planned administration of any of these products during the entire study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to vaccination are eligible. Persons receiving prophylactic antiplatelet medications, e.g., low-dose aspirin, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination. (Subjects suffering from seasonal allergies or asthma under inhalative treatment can be included, as well as subjects with well controlled underlying diseases).
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormalities, as determined by physical examination or laboratory screening tests.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to any constituent of influenza vaccines; or a history of severe adverse reaction to a previous influenza vaccine.
* History of chronic alcohol consumption and/or drug abuse.
* Clinically or virologically confirmed influenza infection within 6 months preceding the study start.
* Any conditions which, in the opinion of the investigator, prevents the subjects from participating in the study.

Min Age: 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2009-09-08; Primary Completion 2009-11-16 (Actual); Study Completion 2010-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Germany (5):
  - GSK Investigational Site, Rednitzhembach, Bavaria
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Peeters M, Regner S, Vaman T, Devaster JM, Rombo L. Safety and immunogenicity of an AS03-adjuvanted A(H1N1)pmd09 vaccine administered simultaneously or sequentially with a seasonal trivalent vaccine in adults 61 years or older: data from two multicentre randomised trials. Vaccine. 2012 Oct 5;30(45):6483-91. doi: 10.1016/j.vaccine.2012.07.081. Epub 2012 Aug 9. PMID 22885014
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113572 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo-Pandemrix-Fluarix Group: Subjects received one dose of placebo intramuscularly in the deltoid region of the dominant arm at Day -21, 2 doses of Pandemrix intramuscularly in the deltoid region of the non-dominant arm at Day 0 and Day 21, and 1 dose of Fluarix intramuscularly in the deltoid region of the dominant arm at Day 42.
- Fluarix-Pandemrix-Placebo Group: Subjects received 1 dose of Fluarix intramuscularly in the deltoid region of the dominant arm at Day -21, 2 doses of Pandemrix intramuscularly in the deltoid of the non-dominant arm at Day 0 and 21, and 1 dose of placebo intramuscularly in the deltoid of the non-dominant arm at Day 42.
Period: Overall Study
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Started | 72 | 73
Completed | 71 | 71
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group | Total
Number analyzed (Participants) | 72 | 73 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.1 (5.16) | 69.7 (5.59) | 69.4 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 34 | 73
  Male | 33 | 39 | 72

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Pandemrix Vaccine Strain
Description: Titers were expressed as GMTs.
  The Pandemrix vaccine strain was A/Cal/7/09.
Time Frame: At Day 42
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for immunogenicity , which included all evaluable subjects for whom immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
titer | 309.8 [246.4 to 389.6] | 227.5 [181.5 to 285.3]

2. Primary Outcome: Number of Subjects With a Titer Greater Than or Equal to 1:10 for Antibodies Against Pandemrix Vaccine Strain
Description: The Pandemrix vaccine strain was A/Cal/7/09.
  The cut-off was a titer of 1:10 and this titer was considered as seropositivity.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
subjects | 64 | 67

3. Primary Outcome: Number of Seroconverted Subjects for Antibodies Against Pandemrix Vaccine Strain
Description: The Pandemrix vaccine strain was A/Cal/7/09.
  A subject seroconverted for haemagglutination inhibition (HI) antibodies was defined as a subject with either a prevaccination (Day 0) HI antibody titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a prevaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
subjects | 61 | 59

4. Primary Outcome: Seroconversion Factor for Antibodies Against Pandemrix Vaccine Strain
Description: Seroconversion Factor (SCF) is defined as the fold increase in serum HI antibody GMTs post-vaccination compared to prevaccination (Day 0).
  The Pandemrix vaccine strain was A/Cal/7/09.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
fold increase | 33.6 [25.5 to 44.3] | 16.5 [12.4 to 21.9]

5. Primary Outcome: Number of Seroprotected Subjects for Antibodies Against Pandemrix Vaccine Strain
Description: The Pandemrix vaccine strain was A/Cal/7/09.
  A seroprotected subject was defined as a subject with a serum HI antibody titer greater than or equal to 1:40.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
subjects | 64 | 67

6. Secondary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Pandemrix Vaccine Strain and Fluarix Vaccine Strains
Description: Pandemrix vaccine strain (A/Cal/7/09) data were assessed up to Month 12. Note that Day 42 data for Pandemrix vaccine strain were already addressed as a primary outcome measure.
  Fluarix vaccine strains (A/Bri/59/07, B/Bri/60/08, and A/Uru/716/07) data were only assessed up to Day 63.
Time Frame: Day -21, Day 0, Day 21, Day 42, Day 63, Month 6 and Month 12
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
titer
  Day -21 A/Cal/7/09 (N=64;67) | 8.7 [6.9 to 11.1] | 7.4 [6.3 to 8.7]
  Day 0 A/Cal/7/09 (N=64;67) | 9.2 [7.3 to 11.7] | 13.8 [11.3 to 16.9]
  Day 21 A/Cal/7/09 (N=64;67) | 147.5 [111.9 to 194.4] | 109.6 [82.4 to 145.8]
  Day 63 A/Cal/7/09 (N=63;66) | 223.8 [181.2 to 276.5] | 174.0 [138.7 to 218.4]
  Month 6 A/Cal/7/09 (N=60;63) | 102.0 [78.6 to 132.3] | 74.1 [59.0 to 92.9]
  Month 12 A/Cal/7/09 (N=60;64) | 35.6 [27.0 to 47.0] | 25.7 [20.8 to 31.9]
  Day -21 A/Bri/59/07 (N=64;67) | 23.1 [18.9 to 28.4] | 20.8 [16.7 to 25.9]
  Day 0 A/Bri/59/07 (N=64;67) | 22.4 [18.2 to 27.5] | 64.0 [50.8 to 80.5]
  Day 42 A/Bri/59/07 (N=64;67) | 32.3 [26.4 to 39.7] | 56.5 [45.3 to 70.5]
  Day 63 A/Bri/59/07 (N=63;66) | 55.7 [45.1 to 68.7] | 49.8 [40.1 to 61.9]
  Day -21 B/Bri/60/08 (N=64;67) | 120.7 [98.7 to 147.7] | 135.6 [107.2 to 171.6]
  Day 0 B/Bri/60/08 (N=64;67) | 118.8 [97.7 to 144.5] | 351.2 [285.6 to 431.9]
  Day 42 B/Bri/60/08 (N=64;67) | 182.2 [154.7 to 214.6] | 291.5 [238.8 to 355.8]
  Day 63 B/Bri/60/08 (N=63;66) | 291.3 [246.2 to 344.7] | 273.3 [225.3 to 331.6]
  Day -21 A/Uru/716/07 (N=64;67) | 26.2 [19.2 to 35.7] | 22.5 [16.2 to 31.2]
  Day 0 A/Uru/716/07 (N=64;67) | 25.5 [18.8 to 34.6] | 100.9 [75.9 to 134.1]
  Day 42 A/Uru/716/07 (N=64;67) | 27.1 [20.7 to 35.4] | 69.2 [51.0 to 93.7]
  Day 63 A/Uru/716/07 (N=63;66) | 85.9 [65.2 to 113.2] | 62.4 [46.9 to 83.2]

7. Secondary Outcome: Number of Subjects With a Titer Greater Than or Equal to 1:10 for Antibodies Against Pandemrix Vaccine Strain and Fluarix Vaccine Strains
Description: The cut-off was a titer of 1:10 and this titer was considered as seropositivity.
  Pandemrix vaccine strain (A/Cal/7/09) data were assessed up to Month 12. Note that Day 42 data for Pandemrix vaccine strain were already addressed as a primary outcome measure.
  Fluarix vaccine strains (A/Bri/59/07, B/Bri/60/08, and A/Uru/716/07) data were only assessed up to Day 63.
Time Frame: At Day -21, Day 0, Day 21, Day 42, Day 63, Month 6 and Month 12
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
subjects
  Day -21 A/Cal/7/09 (N=64;67) | 22 | 21
  Day 0 A/Cal/7/09 (N=64;67) | 26 | 50
  Day 21 A/Cal/7/09 (N=64;67) | 64 | 67
  Day 63 A/Cal/7/09 (N=63;66) | 63 | 66
  Month 6 A/Cal/7/09 (N=60;63) | 60 | 63
  Month 12 A/Cal/7/09 (N=60;64) | 57 | 60
  Day -21 A/Bri/59/07 (N=64;67) | 57 | 58
  Day 0 A/Bri/59/07 (N=64;67) | 56 | 67
  Day 42 A/Bri/59/07 (N=64;67) | 62 | 67
  Day 63 A/Bri/59/07 (N=63;66) | 62 | 66
  Day -21 B/Bri/60/08 (N=64;67) | 64 | 67
  Day 0 B/Bri/60/08 (N=64;67) | 64 | 67
  Day 42 B/Bri/60/08 (N=64;67) | 64 | 67
  Day 63 B/Bri/60/08 (N=63;66) | 63 | 66
  Day -21 A/Uru/716/07 (N=64;67) | 51 | 52
  Day 0 A/Uru/716/07 (N=64;67) | 51 | 66
  Day 42 A/Uru/716/07 (N=64;67) | 57 | 66
  Day 63 A/Uru/716/07 (N=63;66) | 63 | 65

8. Secondary Outcome: Number of Seroconverted Subjects for Antibodies Against Pandemrix Vaccine Strain and Fluarix Vaccine Strains
Description: A seroconverted subject was defined as a subject with either a prevaccination (Day 0) HI antibody titer below 1:10 and a post-vaccination titer greater than or equal to 1:40 or a prevaccination titer greater than or equal to 1:10 and at least a 4-fold increase in post-vaccination titer.
  Pandemrix vaccine strain (A/Cal/7/09) data were generated for Day 21, Month 6 and Month 12.
  Fluarix vaccine strains (A/Bri/59/07, B/Bri/60/08, and A/Uru/716/07) data were generated at 21 days after Fluarix administration, i.e. depending on the group at Day 0 or Day 63 (Day 0/Day 63).
Time Frame: At Day 21, Month 6 and Month 12 for Pandemrix vaccine strain, and at Day 0/Day 63 for Fluarix vaccine strains.
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
subjects
  Day 21 A/Cal/7/09 (N=64;67) | 57 | 43
  Month 6 A/Cal/7/09 (N=60;63) | 48 | 39
  Month 12 A/Cal/7/09 (N=60;64) | 19 | 11
  Day 63/Day 0 A/Bri/56/07 (N=63;67) | 9 | 21
  Day 63/Day 0 B/Bri/60/08 (N=63;67) | 4 | 18
  Day 63/Day 0 A/Uru/716/07 (N=63;67) | 25 | 34

9. Secondary Outcome: Seroconversion Factor for Antibodies Against Pandemrix Vaccine Strain and Fluarix Vaccine Strains
Description: For the definition of seroconversion factor, please refer to the primary outcome measure.
  Pandemrix vaccine strain (A/Cal/7/09) data were generated for Day 21, Month 6 and Month 12.
  Fluarix vaccine strains (A/Bri/59/07, B/Bri/60/08, and A/Uru/716/07) data were generated at 21 days after Fluarix administration, i.e. depending on the group at Day 0 or Day 63 (Day 0/Day 63).
Time Frame: At Day 21, Month 6 and Month 12 for Pandemrix vaccine strain, and at Day 0/Day 63 for Fluarix vaccine strains.
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
fold increase
  Day 21 A/Cal/7/09 (N=64;67) | 16.0 [12.2 to 21.0] | 7.9 [5.8 to 10.8]
  Month 6 A/Cal/7/09 (N=60;63) | 10.9 [8.5 to 14.1] | 5.2 [3.8 to 6.9]
  Month 12 A/Cal/7/09 (N=60;64) | 3.8 [2.9 to 5.0] | 1.8 [1.4 to 2.4]
  Day 63/Day 0 A/Bri/56/07 (N=63;67) | 1.7 [1.4 to 2.1] | 3.1 [2.3 to 4.1]
  Day 63/Day 0 B/Bri/60/08 (N=63;67) | 1.6 [1.4 to 1.8] | 2.6 [2.1 to 3.2]
  Day 63/Day 0 A/Uru/716/07 (N=63;67) | 3.1 [2.5 to 4.0] | 4.5 [3.3 to 6.0]

10. Secondary Outcome: Number of Seroprotected Subjects for Antibodies Against Pandemrix Vaccine Strain and Fluarix Vaccine Strains
Description: A seroprotected subject was defined as a subject with a serum HI antibody titer greater than or equal to 1:40.
  Pandemrix vaccine strain (A/Cal/7/09) data were assessed up to Month 12. Note that Day 42 data for Pandemrix vaccine strain were already addressed as a primary outcome measure.
  Fluarix vaccine strains (A/Bri/59/07, B/Bri/60/08, and A/Uru/716/07) data were only assessed up to Day 63.
Time Frame: Day -21, Day 0, Day 21, Day 42, Day 63, Month 6 and Month 12
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 64 | 67
subjects
  Day -21 A/Cal/7/09 (N=64;67) | 9 | 4
  Day 0 A/Cal/7/09 (N=64;67) | 9 | 12
  Day 21 A/Cal/7/09 (N=64;67) | 60 | 58
  Day 63 A/Cal/7/09 (N=63;66) | 63 | 65
  Month 6 A/Cal/7/09 (N=60;63) | 52 | 53
  Month 12 A/Cal/7/09 (N=60;64) | 28 | 19
  Day -21 A/Bri/59/07 (N=64;67) | 25 | 21
  Day 0 A/Bri/59/07 (N=64;67) | 26 | 50
  Day 42 A/Bri/59/07 (N=64;67) | 30 | 47
  Day 63 A/Bri/59/07 (N=63;66) | 50 | 42
  Day -21 B/Bri/60/08 (N=64;67) | 61 | 63
  Day 0 B/Bri/60/08 (N=64;67) | 61 | 67
  Day 42 B/Bri/60/08 (N=64;67) | 64 | 67
  Day 63 B/Bri/60/08 (N=63;66) | 63 | 66
  Day -21 A/Uru/716/07 (N=64;67) | 30 | 22
  Day 0 A/Uru/716/07 (N=64;67) | 29 | 57
  Day 42 A/Uru/716/07 (N=64;67) | 30 | 47
  Day 63 A/Uru/716/07 (N=63;66) | 54 | 46

11. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms After Administration of Pandemrix
Description: Solicited local symptoms were pain, redness and swelling at the injection site. Solicited general symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating, temperature (defined as axillary temperature equal to or above 37.5 degrees Celsius).
Time Frame: During a 7-Day (Day 0-6) follow-up period after each administration of Pandemrix
Population: The analysis was performed on the Total Vaccinated cohort on subjects with available results
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 72 | 71
subjects
  Pain | 49 | 43
  Redness | 11 | 10
  Swelling | 8 | 11
  Fatigue | 22 | 18
  Headache | 23 | 19
  Joint pain at other location | 20 | 13
  Muscle aches | 23 | 22
  Shivering | 14 | 15
  Sweating | 12 | 13
  Temperature | 2 | 3

12. Secondary Outcome: Number of Subjects With Solicited Local and General Symptoms After Administration of Placebo or Fluarix
Description: Solicited local symptoms were pain, redness and swelling at the injection site. General symptoms were fatigue, headache, joint pain at other location, muscle aches, shivering, sweating, temperature (defined as axillary temperature equal to or above 37.5 degrees Celsius)
Time Frame: During a 7-Day (Day 0-6) follow-up period after each administration of (at Day -21 and at Day 42) placebo or Fluarix
Population: The analysis was performed on the Total Vaccinated cohort on subjects with available results.
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 72 | 72
subjects
  pain Day -21 (N=72;72) | 5 | 12
  redness Day -21 (N=72;72) | 2 | 1
  swelling Day -21 (N=72;72) | 0 | 1
  pain Day 42 (N=69;71) | 17 | 4
  redness Day 42 (N=69;71) | 1 | 0
  swelling Day 42 (N=69;71) | 2 | 0
  fatigue Day -21 (N=72;72) | 9 | 7
  headache Day -21 (N=72;72) | 5 | 10
  joint pain at other location Day -21 (N=72;72) | 7 | 2
  muscle aches Day -21 (N=72;72) | 4 | 6
  shivering Day -21 (N=72;72) | 2 | 4
  sweating Day -21 (N=72;72) | 5 | 6
  temperature Day -21 (N=72;72) | 0 | 1
  fatigue Day 42 (N=69;71) | 10 | 4
  headache Day 42 (N=69;71) | 10 | 8
  joint pain at other location Day 42 (N=69;71) | 8 | 6
  muscle aches Day 42 (N=69;71) | 7 | 5
  shivering Day 42 (N=69;71) | 3 | 3
  sweating Day -21 (N=69;71) | 3 | 4
  temperature Day 42 (N=69;71) | 0 | 0

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Any: any unsolicited AE regardless of intensity or relationship to vaccination. Grade 3: unsolicited AE that prevented normal everyday activity Related: unsolicited AE assessed by the investigator as related to the vaccination
Time Frame: During 21 days (Day 0-20) after each vaccination
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 72 | 73
subjects
  Any | 33 | 37
  Grade 3 | 4 | 10
  Related | 14 | 9

14. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study period (Day 0-364)
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 72 | 73
subjects | 11 | 14

15. Secondary Outcome: Number of Subjects With AEs of Specific Interest
Description: Adverse events of specific interest included auto-immune diseases and other immune mediated disorders.
Time Frame: During the entire study period (Day 0-364)
Population: The analysis was performed on the Total Vaccinated cohort.
Measure: Number; unit: subjects
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Number analyzed (Participants) | 72 | 73
subjects | 0 | 1

ADVERSE EVENTS:
Description: Number of subjects at risk differs for other adverse events, as it depends on the number of subjects with available results. After the different vaccinations there were different numbers of subjects for whom results were available.
Arm/Group | Placebo-Pandemrix-Fluarix Group | Fluarix-Pandemrix-Placebo Group
Serious Adverse Events (participants affected / at risk) | 11/72 | 14/73
Other Adverse Events (participants affected / at risk) | 59/72 | 57/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Pandemrix-Fluarix Group (N=72) | Fluarix-Pandemrix-Placebo Group (N=73)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Sciatica (Nervous system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Death (General disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Eyelid ptosis (Eye disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Femoral arterial stenosis (Vascular disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo-Pandemrix-Fluarix Group (N=72) | Fluarix-Pandemrix-Placebo Group (N=73)
Pain (General disorders) | 49 | 43/71 — after Pandemrix administration
Redness (General disorders) | 11 | 10/71 — after Pandemrix administration
Swelling (General disorders) | 8 | 11/71 — after Pandemrix administration
Pain (General disorders) | 17/69 | 12/72 — after Fluarix administration
Fatigue (General disorders) | 22 | 18/71 — after Pandemrix administration
Headache (General disorders) | 23 | 19/71 — after Pandemrix administration
Joint pain at other location (General disorders) | 20 | 13/71 — after Pandemrix administration
Muscle aches (General disorders) | 23 | 22/71 — after Pandemrix administration
Shivering (General disorders) | 14 | 15/71 — after Pandemrix administration
Sweating (General disorders) | 12 | 13/71 — after Pandemrix administration
Fatigue (General disorders) | 10/69 | 7/72 — after Fluarix administration
Headache (General disorders) | 10/69 | 10/72 — after Fluarix administration
Joint pain at other location (General disorders) | 8/69 | 2/72 — after Fluarix administration
Muscle aches (General disorders) | 7/69 | 6/72 — after Fluarix administration
Shivering (General disorders) | 3/69 | 4/72 — after Fluarix administration
Sweating (General disorders) | 3/69 | 6/72 — after Fluarix administration
Nasopharyngitis (Infections and infestations) | 11 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.